CLINICAL TRIAL: NCT02455882
Title: Tissue Procurement Protocol for Patients Undergoing Treatment for Early-Stage Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: This study was terminated to prevent duplicative research efforts.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Erin Cobain, Clinical Lecturer in Internal Medicine, University of Michigan
Other Study IDs: HUM00084633
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue with invasive disease, blood, and urine samples will be obtained from patients with breast cancer before, during, and after systemic treatment for primary breast cancer and at the time of disease recurrence.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Neoadjuvant: Patients initiating standard of care treatment with primary systemic therapy for breast cancer
- Adjuvant: Patients initiating standard of care treatment with surgery followed by adjuvant chemotherapy for breast cancer
- Recurrence: Patients with a history of breast cancer who are diagnosed with disease recurrence

SUMMARY:
Through the investigators' Breast Care Center at the University of Michigan Comprehensive Cancer Center, the investigators treat approximately 75 patients per year with neoadjuvant chemotherapy. The majority of the remainder of patients with stage II and III disease undergo treatment with adjuvant chemotherapy either on a clinical protocol or as standard of care. There is a subset of women with ER positive disease who do not receive chemotherapy because of favorable tumor characteristics.

This tissue procurement protocol is designed to systematically collect tissue, urine and blood specimens on patients undergoing neoadjuvant systemic therapy or adjuvant chemotherapy, serially following treatment, and/or at the time of disease recurrence in order to investigate mechanisms underlying development of metastatic disease, to identify predictors of response and resistance to therapy, and to test potential new therapies for breast cancer using a combination of patient-derived xenograft creation and new microfluidic technologies.

ELIGIBILITY:
Entry Criteria for patients receiving neoadjuvant or adjuvant therapy (groups 1 and 2)

Inclusion Criteria

* All patients must have a primary invasive breast cancer with the primary tumor intact (T2-4, any N, any M). Inflammatory breast cancer is permitted.
* For the neoadjuvant cohort (group 1), the patient's clinical plan includes neoadjuvant systemic therapy (chemotherapy, hormonal therapy, and/or biologic therapy) prior to surgery on the breast.
* For the adjuvant cohort (group 2), the patient's clinical plan includes surgical resection of the primary breast mass followed by adjuvant chemotherapy (with or without endocrine therapy or biologic therapy such as trastuzumab).
* Patients in the neoadjuvant cohort must have had mammography performed at the University of Michigan, OR outside film review prior to enrollment.
* All patients are required to sign an informed consent document regarding the experimental purpose of the research biopsies and serum banking, in accordance with the University of Michigan IRB standards.

Exclusion Criteria - For the neoadjuvant cohort (group 1): Tumors diagnosed by excisional biopsy, or incisional biopsy that does not leave at least 2 cm of measurable disease by physical examination, mammography, or ultrasound (with the exception of inflammatory breast cancer)

- For the adjuvant cohort (group 2): Tumors diagnosed by excisional or incisional biopsy and which are not likely to have at least 2 cm of residual tumor remaining

* Patients must not have received any prior chemotherapy, hormonal therapy, or radiation therapy for their current breast cancer. Patients who received tamoxifen or other agents for prevention of breast cancer may be included.
* Patients with another active systemic malignancy within the past year.

Entry Criteria for patients with newly diagnosed locoregional or distant disease recurrence (who did not enroll at the time of initial adjuvant or neoadjuvant chemotherapy) (group 3)

Inclusion Criteria

* Patients must have been previously diagnosed with non-invasive or invasive breast cancer.
* Patients must have been diagnosed with biopsy-proven recurrence of breast cancer at any site
* All patients are required to sign an informed consent document regarding the experimental purpose of the research biopsies and serum banking, in accordance with the University of Michigan IRB standards.

Exclusion Criteria

* Patients must not have received any chemotherapy, hormonal therapy, or radiation therapy for treatment of their recurrent breast cancer.
* Patients must not have been diagnosed with another active systemic malignancy within the past year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with newly diagnosed breast cancer or breast cancer recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Collection of samples for analysis of somatic mutations | 5 years
  Mutations in the tumor before and after primary systemic therapy will be examined

SECONDARY OUTCOMES:
Collection of samples for analysis of circulating biomarkers | 5 years
  Change in circulating biomarkers, including extracellular DNA and RNA, over time will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Erin F Cobain, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States